CLINICAL TRIAL: NCT05856890
Title: A Phase 1, Placebo-controlled, Dose-escalation Study of the Safety, Pharmacokinetics, and Antiviral Activity of a Potent Neutralizing Monoclonal Antibody in Individuals With Chronic Hepatitis B Infection
Brief Title: HepB mAb19 in Individuals With Chronic Hepatitis B Infection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Marina Caskey, MD, Professor of Clinical Investigation, Rockefeller University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: RUHBV1; MCA-1037 (Other: Rockefeller University IRB)
Record Dates: First submitted 2023-04-19; First posted 2023-05-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hepatitis b Virus; Hepatitis B
Keywords: monoclonal antibody; HBV; HepB mAb19
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: In Groups 1-4, eligible participants will be randomized at a 3:1 ratio to receive a single intravenous infusion of HepB mAb19 or placebo (normal saline) at one of four increasing dose levels (1 mg/kg, 3 mg/kg, 10 mg/kg and 30 mg/kg). In Group 5 participants will receive HepB mAb19 at the maximum tolerated dose (MTD)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Group 1a: HepB mAb19 1 mg/kg, IV (Experimental): Single intravenous infusion of HepB mAb19, dosed at 1 mg/kg.
  Interventions: Biological: HepB mAb19
- Group 2a: HepB mAb19 3 mg/kg, IV (Experimental): Single intravenous infusion of HepB mAb19, dosed at 3 mg/kg.
  Interventions: Biological: HepB mAb19
- Group 3a: HepB mAb19 10 mg/kg, IV (Experimental): Single intravenous infusion of HepB mAb19, dosed at 10 mg/kg.
  Interventions: Biological: HepB mAb19
- Group 4a: HepB mAb19 30 mg/kg, IV (Experimental): Single intravenous infusion of HepB mAb19, dosed at 30 mg/kg.
  Interventions: Biological: HepB mAb19
- Group 5: Maximum tolerated dose, IV (Experimental): Single intravenous infusion of HepB mAb19, dosed at the MTD
  Interventions: Biological: HepB mAb19
- Group 1b: Placebo 1 mg/kg, IV (Placebo Comparator): Single intravenous infusion of placebo - normal saline, dosed at 1 mg/kg.
  Interventions: Other: Sterile Saline
- Group 2b: Placebo 3 mg/kg, IV (Placebo Comparator): Single intravenous infusion of placebo - normal saline, dosed at 3 mg/kg.
  Interventions: Other: Sterile Saline
- Group 3b: Placebo 10 mg/kg, IV (Placebo Comparator): Single intravenous infusion of placebo - normal saline, dosed at 10 mg/kg.
  Interventions: Other: Sterile Saline
- Group 4b: Placebo 30 mg/kg, IV (Placebo Comparator): Single intravenous infusion of placebo - normal saline, dosed at 30 mg/kg.
  Interventions: Other: Sterile Saline

INTERVENTIONS:
Biological: HepB mAb19 — HepB mAb19 is a human mAb of IgG1kappa isotype that specifically binds to the "a" determinant of the extracellular loop of the HBV surface antigen (HBsAg).
  Arms: Group 1a: HepB mAb19 1 mg/kg, IV; Group 2a: HepB mAb19 3 mg/kg, IV; Group 3a: HepB mAb19 10 mg/kg, IV; Group 4a: HepB mAb19 30 mg/kg, IV; Group 5: Maximum tolerated dose, IV
Other: Sterile Saline — Placebo will be normal sterile saline (NaCl 0.9%).
  Arms: Group 1b: Placebo 1 mg/kg, IV; Group 2b: Placebo 3 mg/kg, IV; Group 3b: Placebo 10 mg/kg, IV; Group 4b: Placebo 30 mg/kg, IV

SUMMARY:
This is a first-in-human, placebo-controlled, single dose, dose-escalation phase 1 study to evaluate the safety, pharmacokinetics and antiviral activity of a highly potent neutralizing anti-HBV monoclonal antibody (mAb), HepB mAb19, which targets the S-protein in individuals with chronic hepatitis B (CHB) on nucleos(t)ide analog therapy (NRTI).

DETAILED DESCRIPTION:
The study has a dose escalation design. In Groups 1-4, eligible participants will be randomized at a 3:1 ratio to receive a single intravenous infusion of HepB mAb19 or placebo (normal saline) at one of four increasing dose levels (1 mg/kg, 3 mg/kg, 10 mg/kg and 30 mg/kg). In Group 5 participants will receive HepB mAb19 at the maximum tolerated dose (MTD). Participants will be followed for 48 weeks after HepB mAb19 or placebo infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70;
* HBV infection confirmed by positive HBsAg for >/= 6 months;
* On HBV-active nucleos(t)ide therapy for >/= 6 months without change in NRTI in the previous 3 months;
* The following laboratory values within 49 days from study entry (day 0):
* HBV DNA below lower limit of quantification;
* HBsAg > 10 IU/mL;
* HBs antibody negative;
* Ability and willingness to provide informed consent;
* For participants who can become pregnant (i.e., participants who have not been post-menopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, or who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy), negative serum or urine pregnancy test at screening and on day 0 (study entry).
* Participants who can become pregnant must agree to use two methods of contraception.
* Partner sterilization with documentation of azoospermia prior to the participant's entry into the study, and this partner is the sole partner for that participant. The documentation of partner sterility can come from the site personnel's review of medical records or medical history interview provided by the participant or the partner. Self-reported documentation of reproductive potential should be entered in the source documents.
* Participants who can impregnate a partner and who are engaging in sexual activity that could lead to pregnancy must agree to use condoms from 10 days prior to study entry and during study follow up to avoid impregnating a partner who can get pregnant.

Exclusion Criteria:

- Clinical symptoms, imaging studies or liver histology suggestive of advanced fibrosis (exclude fibrosis grade 3 and 4 by FibroScan (Fibroscan®< 9 kpa) within 12 months from entry or done at the pre-infusion visit.

Note: If FibroScan results from within 12 months are not available, imaging will be performed at the pre-infusion visit.

* Presence of a LI-RADS4 or 5 liver lesion on imaging within 12 months from entry or done at pre-infusion visit, if prior results not available.
* Alpha fetoprotein > 20 ng/ml Note: AFP above normal but < 20 is acceptable for entry if earlier AFP levels (older than 6 months) are within normal range and imaging is negative in last 3 months).
* HIV-1, HCV or hepatitis delta virus infection within 12 months from entry or done at screen, if prior results not available.
* History of hematopoietic stem cell transplant or solid organ transplant;
* Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, monoclonal antibody or vaccine, or multiple drug allergies (non-active hay fever is acceptable);
* History of cardiovascular disease (e.g., cardiac insufficiency, coronary artery disease, cardiomyopathy, congestive heart failure, family history of congenital long QT syndrome, family history of sudden death);
* History or presence of clinically significant ECG abnormalities based on the average of the triplicate ECG recordings (e.g., QT corrected for heart rate using the Fridericia's correction factor [QTcF] > 450 ms for males and QTcF > 470 ms for females);
* History of systemic corticosteroids, immunosuppressive anti-cancer, systemic interferons or interleukins within the last 6 months;
* History of chronic liver disease from another cause, immune complex disease, or autoimmune diseases that in the opinion of the investigator would preclude participation.
* Any significant acute infection (e.g. influenza, COVID-19) or any other clinically significant illness within 2 weeks prior to Day 0.
* Laboratory abnormalities in the parameters listed below:
* Absolute neutrophil count < 1,000 /mm3
* Hemoglobin < 10 gm/dL
* Platelet count < 150,000 /mm3
* ALT > 2.0 x ULN
* AST > 2.0 x ULN
* Total bilirubin > 1.5 ULN (except individuals with known Gilbert's)
* Albumin < 3.5 gm/dL
* Calculated creatinine clearance < 70 mL/min (using the Cockcroft Gault formula).
* INR >/= 1.2
* Pregnancy or lactation;
* Any vaccination within 14 days prior to IP administration;
* Receipt of anti-HBV mAb therapy of any kind in the past (including HBIG);
* Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate and severity of solicited adverse events that are Grade 2 or above within 2 weeks after administration. | 2 weeks
  The occurrence of solicited AEs will be assessed 2 weeks after IP administration.
Rate and severity of treatment-emerging unsolicited adverse events that are Grade 2 or above (including confirmed laboratory abnormalities) within 2, 12, 24 and 48 weeks after administration. | 48 weeks
  The occurrence of treatment-emerging AEs will be assessed after IP administration
Rate and severity of participants with serious adverse events (SAEs) throughout the study period that are considered related to investigational product and the duration of those SAEs. | 48 weeks
  The occurrence of SAEs will be assessed after IP administration
Rate and severity of participants with potential immune complex disease (ICD) throughout the study period following investigational product (IP) administration. | 48 weeks
  The occurrence of immune complex disease will be assessed after IP administration
Changes in AST within 2,12, 24 and 48 weeks after administration. | 48 weeks
  Changes in AST will be assessed after IP administration
Changes in ALT within 2,12, 24 and 48 weeks after administration | 48 weeks
  Changes in ALT will be assessed after IP administration
Changes in alkaline phosphatase within 2,12, 24 and 48 weeks after administration | 48 weeks
  Changes in alkaline phosphatase will be assessed after IP administration
Changes in bilirubin within 2,12, 24 and 48 weeks after administration | 48 weeks
  Changes in bilirubin will be assessed after IP administration
Changes in albumin within 2,12, 24 and 48 weeks after administration | 48 weeks
  Changes in albumin will be assessed after IP administration
Elimination half-life of HepB mAb19 | 48 weeks
  Elimination half-life (t1/2) will be assessed after IP administration
Clearance (CL/F) of HepB mAb19 | 48 weeks
  Clearance (CL/F) will be assessed after IP administration
Volume of Distribution (Vz/F) of HepB mAb19 | 48 weeks
  Volume of Distribution (Vz/F) will be assessed after IP administration
Area under the curve (AUC) of HepB mAb19 | 48 weeks
  Area under the curve (AUC) will be assessed after IP administration
Decay Curve of HepB mAb19 | 48 weeks
  Decay Curve will be assessed after IP administration

SECONDARY OUTCOMES:
Rate and severity of treatment-related adverse events during study follow up. | 48 weeks
  The occurrence of treatment-related AEs will be assessed after IP administration.
Rate of induced anti-HepB mAb19 antibodies in all study groups. | 48 weeks
  Occurrence of anti-HepB mAb19 antibodies will be assessed at baseline and after IP administration.
Change in quantitative HBsAg levels from baseline (day 0) at each scheduled follow up visit. | 48 weeks
  Serum HBsAg levels will be measured from baseline (day 0) until end of study follow up.
Detection of HBsAg by a qualitative assay at each scheduled follow up visit. | 48 weeks
  Qualitative measure of HBsAg will be performed from baseline (day 0) until end of study follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — The Rockefeller University
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - The Rockefeller University, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Q, Michailidis E, Yu Y, Wang Z, Hurley AM, Oren DA, Mayer CT, Gazumyan A, Liu Z, Zhou Y, Schoofs T, Yao KH, Nieke JP, Wu J, Jiang Q, Zou C, Kabbani M, Quirk C, Oliveira T, Chhosphel K, Zhang Q, Schneider WM, Jahan C, Ying T, Horowitz J, Caskey M, Jankovic M, Robbiani DF, Wen Y, de Jong YP, Rice CM, Nussenzweig MC. A Combination of Human Broadly Neutralizing Antibodies against Hepatitis B Virus HBsAg with Distinct Epitopes Suppresses Escape Mutations. Cell Host Microbe. 2020 Aug 12;28(2):335-349.e6. doi: 10.1016/j.chom.2020.05.010. Epub 2020 Jun 5. PMID 32504577